CLINICAL TRIAL: NCT05574205
Title: The Importance of Dietary Protein Quality for Skeletal Muscle Anabolism in Older Adults
Brief Title: Dietary Protein Quality for Skeletal Muscle Anabolism in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RG_20-157
Record Dates: First submitted 2022-09-29; First posted 2022-10-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia; Dietary Protein; Resistance Exercise
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the high-quality or low-quality condition. Within both conditions single-leg resistance exercise will be undertaken meaning the other non-exercise leg for each participant will act as their own internal control.
Who Masked: Participant
Masking Description: The participant will not know which condition they are under due to the contribution of animal and plant based elements within the diet, the conditions are not immediately obvious. Further, the higher and lower quality supplemental drinks have been made so the taste and texture of which are not discernible.
  The randomisation and counterbalancing will be done by a researcher separate to the project, using anonymised participant codes. The condition participants are under will be also completed before inducting participants. Researchers will be blinded to the condition and which leg was exercised during the analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Quality Protein (Experimental): Participants will consume four high-quality protein containing meals per day (amounting to 1g/kg/day of protein) over a 10-day period. Each meal will contain 75:25 animal:plant protein with most of the animal protein from supplemental high-quality protein powder.
  Interventions: Other: Resistance Exercise; Dietary Supplement: Protein supplementation
- Low Quality Protein (Experimental): Participants will consume four low-quality protein containing meals per day (amounting to 1g/kg/day of protein) over a 10-day period. Each meal will contain 25:75 animal:plant protein with most of the plant protein from supplemental low-quality protein powder.
  Interventions: Other: Resistance Exercise; Dietary Supplement: Protein supplementation

INTERVENTIONS:
Other: Resistance Exercise — Supervised single-leg (unilateral) exercise will be undertaken every other day throughout the dietary intervention
  Other Names: Single-leg resistance exercise
Dietary Supplement: Protein supplementation — Participants will consume a protein supplement alongside a provided diet to control protein amount and quality.

SUMMARY:
Dietary proteins potently augment muscle protein synthesis. Because of poorer anabolic sensitivity with ageing, studies and guidelines recommend higher dietary protein intake for older adults. Although higher doses would benefit skeletal muscle remodelling, large protein consumption is not feasible for many older adults. To circumvent, high-protein quality which possesses a high amino acid profile and digestibility appears to have an emergent role for supporting anabolism. Since currently the best line of defence against age related muscle loss is resistance exercise training and regular protein consumption, emphasising high-quality protein ingestion, such as whey protein, within meals may be feasible and efficacious in supporting musculoskeletal remodelling in older adults, without requirement for large protein doses.

The investigators propose that at low doses, high quality protein will have additive benefit to muscle protein synthesis compared to low-quality protein. Further, combining high-quality protein diets with resistance exercise training will have more profound benefits for muscle protein synthesis and muscle remodelling more so than low-quality protein diets.

DETAILED DESCRIPTION:
Participants will be randomly assigned to a 10-day dietary intervention consuming primarily animal proteins (high-quality condition) or primarily plant proteins (low-quality condition). In both conditions, participants will undertake supervised single-leg resistance exercise training every other day, amassing five days resistance exercise sessions during the study. The groups will aim to be matched and counterbalanced for gender. Equally for unilateral exercise randomisation for leg dominance will aim to be counterbalanced within both groups.

Preliminary assessments:

5 days preceding the start of the dietary intervention, participants will report to the University of Birmingham, Sport, Exercise and Rehabilitation Science for the following:

1. Health questionnaire
2. Written informed consent
3. Anthropometrics (Height and Weight)
4. Body fat (bioelectrical impedance)
5. Start measuring habitual activity (provided with an activity monitor and pedometer)
6. Start measuring habitual diet (provided with diet diary)

2 days preceding the start of the dietary intervention, participants will report to the University of Birmingham, Sport, Exercise and Rehabilitation Science for the following:

1. Saliva sample (participant gives own saliva sample in a tube)
2. 10ml of blood taken for baseline measures (venepuncture by trained phlebotomist)
3. Loading dose of D2O (stable isotope of water ingested in 8 small 50ml doses taken 1 hour apart throughout the day)
4. Find 1 repetition maximum (1RM) during unilateral knee extension.

Dietary intervention each day throughout 10-day intervention participants will provide a saliva sample and then consume a top up dose of D2O, continue wearing an activity tracker and keep a diet diary to record eating times of provided meals.

Meals will be individualised to body weight for each individual to achieve a moderate protein intake of which will then consist of primarily higher quality or lower quality proteins.

Day 0 (first day of diet), participants will report to the University of Birmingham, Sport, Exercise and Rehabilitation Science at 0800h after fasting >10 hours the night prior for the following:

1. Resting metabolic rate (Laying down for 30 minutes to assess gaseous exchange while wearing a mask)
2. Muscle architecture (using non-invasive ultrasonography)
3. Whole-body composition assessment (DXA scan)
4. Bilateral muscle biopsies (small amount of muscle will be taken from the muscle in the thigh (vastus lateralis) by a trained person from the left and right leg, under local anaesthetic)
5. Maximal muscle strength (isometric dynamometry) and neural activation (interpolated twitch) during maximal muscle contraction on both legs in series.
6. Serial blood samples will be taken with a single cannulisation and 8 10ml blood draws taken throughout the visit (before and after consuming a breakfast which is either higher or lower in protein quality, according to the randomised condition).
7. Perceived appetite will be assessed during the visit, before and after breakfast, using visual analogue scales
8. Urine collection tub will be provided to collect urine over the next 24-hours.

After consuming specified breakfast on this visit, participants will continue to eat meals given to them according to their random allocation of either higher or lower quality protein diets.

Day 1, 3, 5, 7, 9

Participants will report to the University of Birmingham, Sport, Exercise and Rehabilitation Science to undergo single-leg resistance exercise on a knee extension machine. Eight sets will be completed on the machine at each visit at 75% of 1RM (determined during preliminary visits and will be supervised).

On day 9, the participant will be given a urine collection tub to collect urine over the next 24-hours.

Day 10 (Diet finishing during this visit), participants will report to the University of Birmingham, Sport, Exercise and Rehabilitation Science at 0800h after fasting >10 hours the night prior for the following assessments:

1. Resting metabolic rate (Laying down for 30 minutes to assess gaseous exchange while wearing a mask)
2. Whole-body composition assessment (DXA scan)
3. Muscle Architecture (using non-invasive ultrasonography)
4. Maximal muscle strength (Isometric Dynamometry) and neural activation during maximal muscle contraction (Interpolated twitch)
5. Bilateral muscle biopsies (small amount of muscle will be taken from the muscle in the thigh (vastus lateralis) from the left and right leg under local anaesthetic
6. Serial blood samples will be taken with a single cannulisation and 8 10ml blood draws taken throughout the visit (before and after consuming the final meal of the diet which is the breakfast which is either higher or lower in protein quality, according to the randomised condition)
7. Perceived appetite will be assessed during the visit, before and after breakfast, using visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged between 50-70 years
* Accustomed to normal physical activity levels (averaging at least 7000 steps a day)
* Healthy body mass (i.e., BMI 18-25 kg/m2)
* General good health indicated by health questionnaire
* Free from COVID-19 (SARS-CoV-2) symptoms.

Exclusion Criteria:

* Habitually high consumers of protein (>1.6g/kg/day) assessed by habitual diet diary
* Food allergies
* Lidocaine allergy
* Smoker
* Bleeding Disorders
* Chronic/systemic illnesses (i.e., renal failure, rheumatoid arthritis, diabetes, poor lung function, heart disease, cancer, uncontrolled hypertension)
* Regular consumption of any analgesic or anti-inflammatory drugs. Taking medications mknown to affect muscle metabolis (e.g. beta-blockers, corticosteroids).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis using muscle biopsies and deuterated water enrichment. | 0-10 days
  Muscle protein synthesis will be assessed during the high-quality and low-quality intervention and compared between exercised and controlled leg.
Leg Strength using dynamometry | 0-10 days
  Evaluating change in leg strength, of trained leg, pre- and post-intervention with high-quality and low-quality protein condition
Neural activation using interpolated twitch | 0-10 days
  Assessing change in neural activation via non-invasive interpolated twitch technique of between exercised legs pre-and post intervention in both protein quality conditions
Muscle architecture using ultrasound | 0-10 days
  Using non-invasive ultrasound to determine change of muscle structure with training between protein quality conditions.

SECONDARY OUTCOMES:
Appetite regulation using questionnaires | 0-10 days (3 hours postprandial)
  Assessing perceived hunger using a validated, 8 question, 100mm visual analogue scales.
Appetite regulation, blood | 0-10 days (3 hours postprandial)
  Assessing the secretion of hunger and appetite hormones within the blood after meals which contain high-quality versus low-quality protein.
Metabolic rate, metabolic cart | 0-10 days
  Evaluating alterations in energy expenditure before and after high-quality or low-quality protein containing meal using a metabolic cart.
Nitrogen balance from urine and dietary protein intake | 0-10 days (24-hour urine collection)
  Evaluating change in nitrogen balance between adhering to high-quality or low-quality protein diets over a 10-day period
Body composition using Duel- energy x-ray absorptiometry (DXA) scan. | 0-10 days
  Change in body composition (muscle mass, fat mass, bone mineral density) will be evaluated using a DXA scanner before and after adhering to single leg resistance exercise paired with either high-quality or low-quality protein diet.
Muscle fibre specific analysis using immunofluorescence microscopy. | 0-10 days
  Evaluate changes in fibre specific differences in the distribution and localisation of key anabolic markers between trained and untrained legs for both protein quality conditions.
Intramuscular signalling using western blotting | 0-10 days
  Evaluate changes in protein content and phosphorylation from the start to the end of the intervention.
Physical activity levels using accelerometery and pedometer | -5-10 days
  Monitoring of habitual and habitual physical activity to evaluate if intensity and duration of activity is similar between habitual and intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, School of Sport, Exercise and Rehabilitation Sciences, Edgbaston, West Midlands, United Kingdom

REFERENCES:
- [Derived] Korzepa M, Quinlan JI, Marshall RN, Rogers LM, Belfield AE, Elhassan YS, Lawson A, Ayre C, Senden JM, Goessens JP, Glover EI, Wallis GA, van Loon LJ, Breen L. Resistance training increases myofibrillar protein synthesis in middle-to-older aged adults consuming a typical diet with no influence of protein source: a randomized controlled trial. Am J Clin Nutr. 2025 Jul;122(1):122-136. doi: 10.1016/j.ajcnut.2025.04.019. Epub 2025 Apr 25. PMID 40288581